CLINICAL TRIAL: NCT00299104
Title: A Randomized, Phase 3, Controlled, Double-Blind, Parallel-Group, Multicenter Study to Evaluate the Safety and Efficacy of Rituximab in Combination With Methotrexate (MTX) Compared to MTX Alone, in Methotrexate-Naive Patients With Active Rheumatoid Arthritis
Brief Title: A Study to Evaluate Rituximab in Combination With Methotrexate in Methotrexate-Naive Patients With Active Rheumatoid Arthritis
Acronym: IMAGE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U3373g; WA17047
Record Dates: First submitted 2006-03-02; First posted 2006-03-06 (Estimated); Results first posted 2011-08-10 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Rituxan; MTX; RA; IMAGE; WA17047
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Folic Acid; Methotrexate; Methylprednisolone; Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Rituximab (0.5 g x 2) + Methotrexate (Experimental): Rituximab intravenously at a dose of 0.5 g on Days 1 and 15 + a background of methotrexate orally at a dose of 7.5 mg escalating by 2.5 mg a week every 1-2 weeks to achieve: 15 mg per week by Week 4 and 20 mg per week by Week 8. Subsequent Rituximab treatment courses were given at 24 week intervals for 5 years provided the Disease Activity Score 28 Joint Count- Erythrocyte Sedimentation Rate (DAS-ESR) result was ≥2.6
  Interventions: Drug: folate; Drug: methotrexate; Drug: methylprednisolone; Drug: rituximab
- Rituximab (1.0 g x 2) + Methotrexate (Experimental): Rituximab intravenously at a dose of 1.0 g on Days 1 and 15 + a background of methotrexate orally at a dose of 7.5 mg escalating by 2.5 mg a week every 1-2 weeks to achieve: 15 mg per week by Week 4 and 20 mg per week by Week 8. Subsequent Rituximab treatment courses were given at 24 week intervals for 5 years provided the Disease Activity Score 28 Joint Count- Erythrocyte Sedimentation Rate (DAS-ESR) result was ≥2.6
  Interventions: Drug: folate; Drug: methotrexate; Drug: methylprednisolone; Drug: rituximab
- Placebo + Methotrexate (Placebo Comparator): Placebo intravenously on Days 1 and 15 + a background of methotrexate orally at a dose of 7.5 mg escalating by 2.5 mg a week every 1-2 weeks to achieve: 15 mg per week by Week 4 and 20 mg per week by Week 8.
  From Week 104 participants were eligible to receive Rituximab 2 X 0.5 g or Rituximab 2 X 1.0 g every 24 weeks.
  Interventions: Drug: folate; Drug: methotrexate; Drug: methylprednisolone; Drug: placebo

INTERVENTIONS:
Drug: folate — Intravenous repeating dose
Drug: methotrexate — Oral or parenteral repeating dose
Drug: methylprednisolone — Intravenous repeating dose
Drug: placebo — Intravenous repeating dose
  Arms: Placebo + Methotrexate
Drug: rituximab — Intravenous repeating dose
  Arms: Rituximab (0.5 g x 2) + Methotrexate; Rituximab (1.0 g x 2) + Methotrexate

SUMMARY:
This is a phase III, randomized, controlled, double-blind, parallel group, international study in approximately 750 patients with active Rheumatoid Arthritis (RA) who are naive to Methotrexate (MTX) therapy. Rheumatoid Factor (RF)-positive and RF-negative patients will be enrolled and will be allocated equally between 3 treatment arms.

ELIGIBILITY:
Inclusion criteria:

* Adult patients 18-80 years of age
* RA for ≥ 2 months;
* Receiving outpatient treatment
* Patients naive to, and considered to be candidates for, methotrexate treatment

Exclusion criteria:

* Rheumatic autoimmune disease other than RA, or significant systemic involvement secondary to RA
* Inflammatory joint disease other than RA, or other systemic autoimmune disorder
* Diagnosis of juvenile rheumatoid arthritis, or RA before the age of 16
* Surgery within 12 weeks of study
* Previous treatment with any approved or investigational biologic agent for RA, an anti-alpha4-integrin antibody or co-stimulation modulator, or cell-depleting therapy
* Concurrent treatment with any biologic agent or DMARD other than methotrexate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 755 (Actual)
Dates: Start 2006-01; Primary Completion 2008-09 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arndt Schottelius, M.D., Study Director — Genentech, Inc.

REFERENCES:
- [Derived] Tak PP, Rigby W, Rubbert-Roth A, Peterfy C, van Vollenhoven RF, Stohl W, Healy E, Hessey E, Reynard M, Shaw T. Sustained inhibition of progressive joint damage with rituximab plus methotrexate in early active rheumatoid arthritis: 2-year results from the randomised controlled trial IMAGE. Ann Rheum Dis. 2012 Mar;71(3):351-7. doi: 10.1136/annrheumdis-2011-200170. Epub 2011 Oct 19. PMID 22012969
- [Derived] Rigby W, Ferraccioli G, Greenwald M, Zazueta-Montiel B, Fleischmann R, Wassenberg S, Ogale S, Armstrong G, Jahreis A, Burke L, Mela C, Chen A. Effect of rituximab on physical function and quality of life in patients with rheumatoid arthritis previously untreated with methotrexate. Arthritis Care Res (Hoboken). 2011 May;63(5):711-20. doi: 10.1002/acr.20419. PMID 21557525
- [Derived] Tak PP, Rigby WF, Rubbert-Roth A, Peterfy CG, van Vollenhoven RF, Stohl W, Hessey E, Chen A, Tyrrell H, Shaw TM; IMAGE Investigators. Inhibition of joint damage and improved clinical outcomes with rituximab plus methotrexate in early active rheumatoid arthritis: the IMAGE trial. Ann Rheum Dis. 2011 Jan;70(1):39-46. doi: 10.1136/ard.2010.137703. Epub 2010 Oct 11. PMID 20937671

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Started | 251 | 252 | 252
Safety/ITT: Received Study Drug | 249 | 249 | 250
Completed Week 24 | 227 | 240 | 241
Completed Week 52 | 213 | 227 | 232
Completed Week 104 | 178 | 213 | 216
Completed | 62 (Completed Week 152) | 77 | 80
Not Completed | 189 | 175 | 172
Not completed — Adverse Event | 14 | 9 | 7
Not completed — Death | 1 | 1 | 1
Not completed — Insufficient therapeutic response | 34 | 13 | 8
Not completed — Failure to return | 9 | 8 | 8
Not completed — Violation of selection criteria | 1 | 2 | 0
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Refused treatment | 9 | 2 | 2
Not completed — Withdrew consent | 14 | 19 | 9
Not completed — Administrative reasons | 106 | 120 | 137
Period: Safety Follow-Up (SFU) Period
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Started | 184 (All participants who received treatment were to enter SFU even if withdrawn during treatment period.) | 212 (All participants who received treatment were to enter SFU even if withdrawn during treatment period.) | 213 (All participants who received treatment were to enter SFU even if withdrawn during treatment period.)
Completed | 129 | 171 | 176
Not Completed | 55 | 41 | 37
Not completed — Death | 3 | 2 | 1
Not completed — Lost to Follow-up | 9 | 11 | 20
Not completed — Withdrawal by Subject | 16 | 21 | 11
Not completed — Administrative reasons | 27 | 7 | 5
Period: Extended Safety Follow-Up (ESFU) Period
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Started | 34 (Only participants with CD19+ B-cell counts below baseline level or less than 80 cells/microliter.) | 40 (Only participants with CD19+ B-cell counts below baseline level or less than 80 cells/microliter.) | 51 (Only participants with CD19+ B-cell counts below baseline level or less than 80 cells/microliter.)
Completed | 29 | 31 | 39
Not Completed | 5 | 9 | 12
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 2 | 2 | 2
Not completed — Withdrawal by Subject | 2 | 4 | 8
Not completed — Administrative reasons | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate | Total
Number analyzed (Participants) | 249 | 249 | 250 | 748
Age, Continuous [Mean (Standard Deviation); unit: years] — Intent-to-treat population
  years | 48.06 (12.692) | 47.87 (13.391) | 47.89 (13.324) | 47.94 (13.136)
Sex: Female, Male [Count of Participants; unit: Participants] — Intent-to-treat population
  Participants
    Female | 192 | 203 | 212 | 607
    Male | 57 | 46 | 38 | 141

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Modified Total Sharp Score (mTSS) From Screening at Week 52
Description: Rate of progression in structural joint damage (PJD) by change in Total Modified Sharp Score (TMSS) from screening to Week 52 in the modified intent-to-treat (MITT) population. TMSS is the sum of the erosion score (ES) and the joint space narrowing (JSN) score and has a range of 0 to 398. The ES is the sum of joint scores collected for 46 joints and has a range of 0 to 230. The JSN is the sum of joint scores collected for 42 joints and has a range of 0 to 168. A score of 0 would indicate no change and higher scores represent a worsening of joint erosions and joint space narrowing.
Time Frame: Baseline and week 52
Population: Modified intent-to-treat population includes patients with a screening and at least one post-baseline radiographic evaluation, grouped as randomized. Linear interpolation/extrapolation used for missing data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Number analyzed (Participants) | 232 | 239 | 244
Score on a scale | 1.079 (4.0934) | 0.646 (1.9196) | 0.359 (1.0095)
Statistical Analysis 1: Comparison: Placebo + Methotrexate vs Rituximab (0.5 g x 2) + Methotrexate vs Rituximab (1.0 g x 2) + Methotrexate; Comparing all three treatment groups; Test type: Superiority or Other; p = 0.0016, Kruskal-Wallis — The Closure Principle was used to adjust for multiple comparisons
Statistical Analysis 2: Comparison: Placebo + Methotrexate vs Rituximab (0.5 g x 2) + Methotrexate; Rituximab 2 x 0.5 g + Methotrexate arm versus Placebo + Methotrexate, stratified for region and baseline rheumatoid factor (RF) status; Test type: Superiority or Other; p = 0.1824, Van-Elteren — The Closure Principle was used to adjust for multiple comparisons
Statistical Analysis 3: Comparison: Placebo + Methotrexate vs Rituximab (1.0 g x 2) + Methotrexate; Rituximab 2 x 1.0 g + Methotrexate arm versus Placebo + Methotrexate, stratified for region and baseline RF status; Test type: Superiority or Other; p = 0.0004, Van-Elteren — The Closure Principle was used to adjust for multiple comparisons

2. Secondary Outcome: Change From Baseline in Modified Sharp Erosion Score at Week 52
Description: Rate of progression in structural joint damage (PJD) by change in modified Sharp erosion score from screening to Week 52. The ES is the sum of joint scores collected for 46 joints and has a range of 0 to 230. A score of 0 would indicate no change and higher scores represent a worsening of joint erosions.
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Number analyzed (Participants) | 232 | 239 | 244
Score on a scale | 0.738 (2.0480) | 0.453 (1.2065) | 0.233 (0.6252)
Statistical Analysis 1: Comparison: Placebo + Methotrexate vs Rituximab (0.5 g x 2) + Methotrexate vs Rituximab (1.0 g x 2) + Methotrexate; Comparing all three treatment groups; Test type: Superiority or Other; p = 0.0004, Kruskal-Wallis — The Closure Principle was used to adjust for multiple comparisons. This was a secondary endpoint in a hierarchical testing structure
Statistical Analysis 2: Comparison: Placebo + Methotrexate vs Rituximab (0.5 g x 2) + Methotrexate; Rituximab 2 x 0.5 g + Methotrexate versus Placebo + Methotrexate, stratified for region and baseline RF status; Test type: Superiority or Other; p = 0.1194, Van-Elteren — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Placebo + Methotrexate vs Rituximab (1.0 g x 2) + Methotrexate; Rituximab 2 x 1.0 g + Methotrexate versus Placebo + Methotrexate, stratified for region and baseline RF status; Test type: Superiority or Other; p = 0.0001, Van-Elteren — [p-value comment as in outcome 2, analysis 1]

3. Secondary Outcome: Percentage of Patients Without Radiographic Progression at Week 52
Description: Percentage of patients without radiographic progression at Week 52, defined as change in total modified Sharp score (TMSS) <= 0. TMSS is the sum of the erosion score (ES) and the joint space narrowing (JSN) score and has a range of 0 to 398. The ES is the sum of joint scores collected for 46 joints and has a range of 0 to 230. The JSN is the sum of joint scores collected for 42 joints and has a range of 0 to 168. A score of 0 would indicate no change.
Time Frame: Baseline, Week 52
Population: Modified intent-to-treat population includes patients with a screening and at least one post-baseline radiographic evaluation, grouped as randomized. Patients with missing data are classified as progressing.
Measure: Number; unit: Percentage
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Number analyzed (Participants) | 232 | 239 | 244
Percentage | 53.4 | 57.7 | 63.5
Statistical Analysis 1: Comparison: Placebo + Methotrexate vs Rituximab (0.5 g x 2) + Methotrexate; Rituximab 2 x 0.5 g + Methotrexate arm versus Placebo + Methotrexate, stratified for region and baseline RF status; Test type: Superiority or Other; p = 0.3803, Cochran-Mantel-Haenszel — This was a secondary endpoint in a hierarchical testing structure; Mean Difference (Net) = 0.04, 95% CI [-0.05 to 0.13]
Statistical Analysis 2: Comparison: Placebo + Methotrexate vs Rituximab (1.0 g x 2) + Methotrexate; Rituximab 2 x 1.0 g + Methotrexate arm versus Placebo + Methotrexate, stratified for region and baseline RF status; Test type: Superiority or Other; p = 0.0309, Cochran-Mantel-Haenszel — This was a secondary endpoint in a hierarchical testing structure; Mean Difference (Net) = 0.10, 95% CI [0.01 to 0.18]

4. Secondary Outcome: Percentage of Patients Without Radiographic Progression in Total Erosion Score at Week 52
Description: No radiographic progression is defined as a change in the total erosion score at Week 52 of less than or equal to zero.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Number analyzed (Participants) | 232 | 239 | 244
Percentage of Participants | 54.7 | 59.0 | 66.8
Statistical Analysis 1: Comparison: Placebo + Methotrexate vs Rituximab (0.5 g x 2) + Methotrexate; Rituximab (0.5 g x 2) + Methotrexate versus Placebo + Methotrexate, stratified for region and baseline RF status; Test type: Superiority or Other; p = 0.3752, Cochran-Mantel-Haenszel — This was a secondary endpoint in a hierarchical testing structure
Statistical Analysis 2: Comparison: Placebo + Methotrexate vs Rituximab (1.0 g x 2) + Methotrexate; Rituximab (1.0 g x 2) + Methotrexate verus Placebo + Methotrexate, stratified for region and Baseline RF status; Test type: Superiority or Other; p = 0.0081, Cochran-Mantel-Haenszel — This was a secondary endpoint in a hierarchical testing structure

5. Secondary Outcome: Change From Baseline in Modified Joint Space Narrowing (JSN) Score at Week 52
Description: Rate of progression in structural joint damage (PJD) by change in modified joint space narrowing (JSN) from screening to Week 52. The JSN is the sum of joint scores collected for 42 joints and has a range of 0 to 168. A score of 0 would indicate no change and higher scores represent a worsening of joint space narrowing.
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Number analyzed (Participants) | 232 | 239 | 244
Score on a scale | 0.341 (2.2408) | 0.193 (0.9422) | 0.126 (0.6363)
Statistical Analysis 1: Comparison: Placebo + Methotrexate vs Rituximab (0.5 g x 2) + Methotrexate vs Rituximab (1.0 g x 2) + Methotrexate; Comparing all three treatment groups; Test type: Superiority or Other; p = 0.5939, Kruskal-Wallis — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo + Methotrexate vs Rituximab (0.5 g x 2) + Methotrexate; Rituximab 2 x 0.5 g + Methotrexate arm versus Placebo + Methotrexate, stratified for region and baseline RF status; Test type: Superiority or Other; p = 0.5478, Van-Elteren — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Placebo + Methotrexate vs Rituximab (1.0 g x 2) + Methotrexate; Rituximab 2 x 1.0 g + Methotrexate arm versus Placebo + Methotrexate, stratified for region and baseline RF status; Test type: Superiority or Other; p = 0.3096, Van-Elteren — [p-value comment as in outcome 2, analysis 1]

6. Secondary Outcome: Change From Baseline in the Modified Total Sharp Score at Week 24
Description: The modified total sharp score is the sum of the erosion score (ES) and the joint space narrowing (JSN) score and has a range of 0 to 398. The ES is the sum of joint scores collected for 46 joints and has a range of 0 to 230. The JSN is the sum of joint scores collected for 42 joints and has a range of 0 to 168. A score of 0 would indicate no change and higher scores represent a worsening of joint erosions and joint space narrowing.
Time Frame: Baseline, Week 24
Population: Participants from the Modified Intent to Treat (MITT) population includes all randomized participants who received at least one infusion and had both screening and post-baseline radiographic assessments at the given time point for analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Number analyzed (Participants) | 226 | 238 | 242
Score on a scale | 0.701 (2.9116) | 0.508 (1.7349) | 0.328 (0.9443)

7. Secondary Outcome: Change From Baseline in the Total Erosion Score at Week 24
Description: Total Erosion Score is determined by evaluation of fourteen sites in each wrist and hand and six joints in each foot using an eight-point scale from 0 (normal: no erosions) to 3.5 (Very severe; erosions of 100% of the articular surfaces. The Total Erosion Score at Week 24 - Total Erosion Score at baseline is calculated.
Time Frame: Baseline, Week 24
Population: Participants from the modified intent-to-treat population (includes patients with a screening and at least one post-baseline radiographic evaluation, grouped as randomized) who had data available at Week 24 for analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Number analyzed (Participants) | 226 | 238 | 242
Score on a scale | 0.491 (1.3789) | 0.404 (1.0390) | 0.220 (0.5802)

8. Secondary Outcome: Change From Baseline in Modified Joint Space Narrowing (JSN) Score at Week 24
Description: Joint Space Narrowing is the sum of joint scores collected for 42 joints and has a range of 0 to 168. A score of 0 would indicate no change and higher scores represent a worsening of joint space narrowing.
Time Frame: Baseline, Week 24
Population: Participants from the modified intent-to-treat population (includes patients with a screening and at least one post-baseline radiographic evaluation, grouped as randomized) with data available at Week 24 for analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Number analyzed (Participants) | 226 | 238 | 242
Score on a scale | 0.210 (1.7403) | 0.176 (0.8949) | 0.108 (0.6118)

9. Secondary Outcome: Percentage of Participants Without Radiographic Progression at Week 24
Description: Percentage of patients without radiographic progression at Week 24 defined as change in total modified Sharp score (TMSS) ≤ 0. TMSS is the sum of the erosion score (ES) and the joint space narrowing (JSN) score and has a range of 0 to 398. The ES is the sum of joint scores collected for 46 joints and has a range of 0 to 230. The JSN is the sum of joint scores collected for 42 joints and has a range of 0 to 168. A score of 0 would indicate no change.
Time Frame: Baseline, Week 24
Population: Modified Intent to Treat (MITT) population includes all randomized participants who received at least one infusion and had both screening and post-baseline radiographic assessments. Patients with missing data are classified as progressing
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Number analyzed (Participants) | 233 | 239 | 244
Percentage of Participants | 59.7 | 65.3 | 71.7

10. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR) ACR50 Response at Week 52
Description: To achieve an ACR50 response requires at least a 50% improvement compared with baseline in both Total Joint Count and Swollen Joint Count, as well as a 50% improvement in three of five additional measurements from:
  * the physician's global assessment of disease activity
  * patient's global assessment of disease activity
  * patient's assessment of pain
  * HAQ-DI (Health Assessment Questionnaire disability index)
  * an acute phase reactant C-Reactive Protein (CRP). (If CRP was missing then Erythrocyte Sedimentation Rate (ESR) was used if available.)
Time Frame: Week 52
Population: Intent to treat (ITT) population includes all randomized participants who received at least one infusion. Patients are considered non-responders if data are missing or from the point of withdrawal, rescue use or receipt of non-permitted Disease-modifying anti-rheumatic drugs (DMARDs).
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Number analyzed (Participants) | 249 | 249 | 250
Percentage of Participants | 41.8 | 59.4 | 64.8
Statistical Analysis 1: Comparison: Placebo + Methotrexate vs Rituximab (0.5 g x 2) + Methotrexate; Rituximab 2 x 0.5 g + Methotrexate arm versus Placebo + Methotrexate, stratified for region and baseline RF status; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — This was a secondary endpoint in a hierarchical testing structure
Statistical Analysis 2: Comparison: Placebo + Methotrexate vs Rituximab (1.0 g x 2) + Methotrexate; Rituximab 2 x 1.0 g + Methotrexate arm versus Placebo + Methotrexate, stratified for region and baseline RF status; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — This was a secondary endpoint in a hierarchical testing structure

11. Secondary Outcome: Change From Baseline in the Disease Activity Score 28 Joint Count- Erythrocyte Sedimentation Rate (DAS28-ESR) at Week 52
Description: DAS28-ESR is calculated from the following formula:
  (0.56 * TJC) + (0.28 * SJC) + (0.70 * ln ESR) + (0.014 * GH) TJC = tender joint count, based on 28 joints SJC = swollen joint count, based on 28 joints ESR = erythrocyte sedimentation rate in mm/h GH = patient's global assessment of disease activity A DAS28-ESR score of 5.1 or above is considered to indicate high disease activity. Patients can also be defined as having low disease activity (DAS28-ESR ≤ 3.2) or remission (DAS28-ESR < 2.6).
Time Frame: Baseline, Week 52
Population: Participants from the Intent to treat (ITT) population includes all randomized participants who received at least one infusion who had data available for analyses. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Number analyzed (Participants) | 244 | 247 | 248
Score on a scale | -2.33 (1.691) | -3.35 (1.663) | -3.46 (1.640)

12. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR) ACR70 Response at Week 52
Description: To achieve an ACR70 response requires at least a 70% improvement compared with baseline in both Total Joint Count and Swollen Joint Count, as well as a 70% improvement in three of five additional measurements from:
  * the physician's global assessment of disease activity
  * patient's global assessment of disease activity
  * patient's assessment of pain
  * HAQ-DI (Health Assessment Questionnaire disability index)
  * an acute phase reactant C-Reactive Protein (CRP). (If CRP was missing then Erythrocyte Sedimentation Rate (ESR) was used if available.)
Time Frame: Baseline, Week 52
Population: as for outcome 10
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Number analyzed (Participants) | 249 | 249 | 250
Percentage of Participants | 24.9 | 42.2 | 46.8

13. Secondary Outcome: Percentage of Participants With DAS28-ESR Remission at Week 52
Description: The DAS28-4(ESR) score is a measure of the subject's disease activity. It is based on the tender joint count (28 joints), swollen joint count (28 joints), patient's global assessment of disease activity (mm), and ESR. DAS28-4(ESR) scores range from 0 - 10.
  Remission is defined as achieving a DAS28-ESR score of less than 2.6
Time Frame: Week 52
Population: Participants from the Intent to treat (ITT) population includes all randomized participants who received at least one infusion with data available for analyses.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Number analyzed (Participants) | 247 | 248 | 249
Percentage of Participants | 12.6 | 25.4 | 30.5

14. Secondary Outcome: Percentage of Participants With European League Against Rheumatism (EULAR) Good Response at Week 52
Description: European League Against Rheumatism (EULAR) criteria reflects an improvement in disease activity and an attainment of a lower degree of disease activity. A good response is defined as an improvement in the DAS28-ESR of > 1.2 compared with baseline, and attainment of a DAS28-ESR of < 3.2.
Time Frame: Baseline, Week 52
Population: Intent to treat (ITT) population includes all randomized participants who received at least one infusion. Patients are considered non-responders if data are missing
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Number analyzed (Participants) | 249 | 249 | 250
Percentage of Participants | 18.1 | 39.0 | 41.6

15. Secondary Outcome: The Percentage of Participants With Major Clinical Response at Week 52
Description: Major clinical response is defined as a continuous six-month period of success by the ACR70.
  ACR70= 70% improvement compared with baseline in both Total Joint Count and Swollen Joint Count, as well as a 70% improvement in 3 of five additional measurements from:
  * the physician's global assessment of disease activity
  * patient's global assessment of disease activity
  * patient's assessment of pain
  * HAQ-DI (Health Assessment Questionnaire disability index)
  * an acute phase reactant C-Reactive Protein (CRP). (If CRP was missing then Erythrocyte Sedimentation Rate (ESR) was used if available.)
Time Frame: Week 52
Population: Intent to treat (ITT) population includes all randomized participants who received at least one infusion.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Number analyzed (Participants) | 249 | 249 | 250
Percentage of Participants | 8.4 | 18.1 | 21.2

16. Secondary Outcome: Percentage of Participants With DAS28-ESR Low Disease Activity at Week 52
Description: The DAS28-4(ESR) score is a measure of the subject's disease activity. It is based on the tender joint count (28 joints), swollen joint count (28 joints), patient's global assessment of disease activity (mm), and ESR. DAS28-4(ESR) scores range from 0 - 10.
  Low disease activity is defined as achieving a DAS28-ESR score of less than or equal to 3.2
Time Frame: Week 52
Population: Participants from the Intent to treat (ITT) population includes all randomized participants who received at least one infusion who had data available for analyses.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Number analyzed (Participants) | 247 | 248 | 249
Percentage of Participants | 19.8 | 40.3 | 43.0

17. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR) ACR20 Response at Week 52
Description: To achieve an ACR20 response requires at least a 20% improvement compared with baseline in both Total Joint Count and Swollen Joint Count, as well as a 20% improvement in three of five additional measurements from:
  * the physician's global assessment of disease activity
  * patient's global assessment of disease activity
  * patient's assessment of pain
  * HAQ-DI (Health Assessment Questionnaire disability index)
  * an acute phase reactant C-Reactive Protein (CRP). (If CRP was missing then Erythrocyte Sedimentation Rate (ESR) was used if available.)
Time Frame: Baseline, Week 52
Population: as for outcome 10
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Number analyzed (Participants) | 249 | 249 | 250
Percentage of Participants | 64.3 | 76.7 | 80.0

18. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR) ACR90 Response at Week 52
Description: To achieve an ACR90 response requires at least a 90% improvement compared with baseline in both Total Joint Count and Swollen Joint Count, as well as a 90% improvement in three of five additional measurements from:
  * the physician's global assessment of disease activity
  * patient's global assessment of disease activity
  * patient's assessment of pain
  * HAQ-DI (Health Assessment Questionnaire disability index)
  * an acute phase reactant C-Reactive Protein (CRP). (If CRP was missing then Erythrocyte Sedimentation Rate (ESR) was used if available.)
Time Frame: Baseline, Week 52
Population: as for outcome 10
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Number analyzed (Participants) | 249 | 249 | 250
Percentage of Participants | 9.2 | 17.3 | 16.4

19. Secondary Outcome: Change in Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F) Score From Baseline at Week 52
Description: FACIT-F is a 13-item questionnaire. Patients scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the patient's response to the questions (with the exception of 2 negatively stated), the greater the patient's fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the patient's response). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score). A higher score reflects an improvement in the patient's health status.
Time Frame: Baseline, Week 52
Population: Participants from the Intent to treat (ITT) population includes all randomized participants who received at least one infusion who had data available for analyses. Observed data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Number analyzed (Participants) | 198 | 206 | 218
Score on a scale | 10.154 (11.1344) | 11.833 (11.5807) | 12.426 (12.2535)

20. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Week 52
Description: The Stanford Health Assessment Questionnaire disability index (HAQ-DI) is a patient completed questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip,and common daily activities. Each domain has at least two component questions. There are four possible responses for each component ranging from 0(without any difficulty) to 4 (unable to do).HAQ-DI=sum of worst scores in each domain divided by the number of domains answered. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 52
Population: Intent-to treat Population includes all randomized participants who received at least one dose of study drug. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Number analyzed (Participants) | 248 | 247 | 249
Score on a scale | -0.800 (0.7764) | -1.038 (0.7625) | -1.023 (0.7634)
Statistical Analysis 1: Comparison: Placebo + Methotrexate vs Rituximab (0.5 g x 2) + Methotrexate; Rituximab (0.5 g x 2) + Methotrexate versus Placebo + Methotrexate stratified for region and RF status; Test type: Superiority or Other; p < 0.0001, ANOVA — Secondary endpoint in hierarchical testing structure
Statistical Analysis 2: Comparison: Placebo + Methotrexate vs Rituximab (1.0 g x 2) + Methotrexate; Rituximab (1.0 g x 2) + Methotrexate versus Placebo + Methotrexate, stratified for region and baseline RF status; Test type: Superiority or Other; p < 0.0001, ANOVA — Secondary endpoint in hierarchical testing structure

21. Secondary Outcome: Change From Baseline in the SF-36 Physical Health Component Summary Score at Week 52 and Week 104
Description: The SF-36 is a questionnaire used to assess physical functioning and is made up of eight domains: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional and Mental Health. Transforming and standardizing these domains leads to the calculation of the Physical (PCS) and Mental (MCS) Component Summary measures. Scores ranging from 0 to 100, with 0=worst score (or quality of life) and 100=best score. A positive change from baseline indicates improvement.
  Means are adjusted for baseline value, Rheumatoid Factor status and region.
Time Frame: Baseline, Week 52, Week 104
Population: Intent to treat (ITT) population includes all participants who received at least one infusion. Last observation carried forward. "n" in each of the categories is the number of participants with data available for analyses at the given time point.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Number analyzed (Participants) | 249 | 249 | 250
Score on a scale
  Week 52 (n=239,236,241) | 8.953 (9.3986) | 11.022 (9.6246) [-0.331 to 3.504] | 12.205 (9.4986) [1.214 to 5.026]
  Week 104 (n=240,236,242) | 8.617 (9.8500) | 11.032 (9.9631) [1.590 to 4.787] | 12.649 (10.4331) [2.749 to 5.920]

22. Secondary Outcome: Change From Baseline in the SF-36 Mental Health Component Summary Score at Week 52 and Week 104
Description: as for outcome 21
Time Frame: Baseline, Weeks 52, Week 104
Population: Intent to treat (ITT) population includes all randomized participants who received at least one infusion. Last observation carried forward. "n" in each of the categories is the number of participants with data available for analyses at the given time point.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Number analyzed (Participants) | 249 | 249 | 250
Score on a scale
  Week 52 (n=239,236,241) | 6.689 (13.1160) | 7.718 (11.8903) | 8.167 (12.1709)
  Week 104 (n= 240,236,242) | 6.295 (13.9813) | 7.617 (12.0793) | 9.066 (12.5325)

23. Secondary Outcome: Percentage of Participants With Categorical Change in Health Assessment Questionnaire- Disability Index (HAQ-DI) From Baseline at Week 52
Description: The Stanford Health Assessment Questionnaire disability index (HAQ-DI) is a patient completed questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and common daily activities. Each domain has at least two component questions. There are four possible responses for each component on a scale of 0 (without difficulty) to 3 (unable to do). Higher scores=greater dysfunction.
  Improved:HAQ-DI score change <=-0.22 Unchanged:HAQ-DI score change -0.22 to 0.22 Worsened:HAQ score => 0.22
Time Frame: Baseline, Week 52
Population: Intent to treat (ITT) population includes all randomized participants who received at least one infusion. Last observation carried forward.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Number analyzed (Participants) | 249 | 249 | 250
Percentage of participants
  Improved | 77.1 | 86.7 | 86.8
  Unchanged | 14.1 | 8.8 | 8.0
  Worsened | 8.4 | 3.6 | 4.4
  Not Assessable | 0.4 | 0.8 | 0.8

24. Secondary Outcome: Percentage of Patients With Minimally Clinically Important Difference (MCID) in the SF-36 Physical Health Component Score at Week 52
Description: MCID is defined as a change from baseline in SF-36 Physical Health Component Score of >5.42.
  SF-36 is a questionnaire used to assess physical functioning and is made up of eight domains: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional and Mental Health. Transforming and standardizing these domains leads to the calculation of the Physical (PCS) and Mental (MCS) Component Summary measures. Scores ranging from 0 to 100, with 0=worst score (or quality of life) and 100=best score. A positive change from baseline indicates improvement.
Time Frame: Baseline, Week 52
Population: Participants from the Intent-to-treat population, includes all randomized participants who received at least one dose of study drug, with data available for analysis at Baseline and Week 52. Last observation carried forward.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Number analyzed (Participants) | 239 | 236 | 242
Percentage of Participants | 63.2 | 69.9 | 76.4

25. Secondary Outcome: Percentage of Patients With Minimally Clinically Important Difference (MCID) in the SF-36 Mental Health Component Score at Week 52
Description: MCID is defined as a change from baseline in SF-36 Mental Health Component Score of >6.33.
  SF-36 is a questionnaire used to assess physical functioning and is made up of eight domains: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional and Mental Health. Transforming and standardizing these domains leads to the calculation of the Physical (PCS) and Mental (MCS) Component Summary measures. Scores ranging from 0 to 100, with 0=worst score (or quality of life) and 100=best score. A positive change from baseline indicates improvement.
Time Frame: Baseline, Week 52
Population: as for outcome 24
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Number analyzed (Participants) | 239 | 236 | 242
Percentage of Participants | 49.0 | 50.8 | 57.0

26. Secondary Outcome: Change From Baseline in the Modified Total Sharp Score at Week 104
Description: as for outcome 6
Time Frame: Baseline, Week 104
Population: Participants from the Modified Intent to Treat (MITT) population includes all randomized participants who received at least one infusion and had both screening and post-baseline radiographic assessments at the given time-point for analysis. Linear extrapolation was used for missing data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Number analyzed (Participants) | 229 | 238 | 243
Score on a scale | 1.948 (5.5782) | 0.761 (2.6181) | 0.406 (1.4312)
Statistical Analysis 1: Comparison: Placebo + Methotrexate vs Rituximab (1.0 g x 2) + Methotrexate; Week 104: Rituximab 2 x 0.5 g + Methotrexate arm versus Placebo + Methotrexate, stratified for region and baseline rheumatoid factor (RF) status; Test type: Superiority or Other; p < 0.0001, Van-Elteren — This was a secondary endpoint in a hierarchical testing structure

27. Secondary Outcome: Change From Baseline in the Total Erosion Score at Week 104
Description: Total Erosion Score is determined by evaluation of fourteen sites in each wrist and hand and six joints in each foot using an eight-point scale from 0 (normal: no erosions) to 3.5 (Very severe; erosions of 100% of the articular surfaces. The change from the score at baseline to week 104 is calculated.
Time Frame: Baseline, Week 104
Population: Participants from the Modified Intent to Treat (MITT) population includes all randomized participants who received at least one infusion and who had both screening and post-baseline radiographic assessments at the given time point for analyses. Linear extrapolation used for missing data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Number analyzed (Participants) | 229 | 238 | 243
Score on a scale | 1.315 (3.2466) | 0.499 (1.7221) | 0.227 (0.7939)

28. Secondary Outcome: Percentage of Participants Without Radiographic Progression at Week 104
Description: Percentage of patients without radiographic progression at Week 104, defined as change in total modified Sharp score (TMSS) ≤ 0. TMSS is the sum of the erosion score (ES) and the joint space narrowing (JSN) score and has a range of 0 to 398. The ES is the sum of joint scores collected for 46 joints and has a range of 0 to 230. The JSN is the sum of joint scores collected for 42 joints and has a range of 0 to 168. A score of 0 would indicate no change.
Time Frame: Baseline, Week 104
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Number analyzed (Participants) | 233 | 239 | 244
Percentage of Participants | 37.3 | 49.4 | 56.6

29. Secondary Outcome: Percentage of Participants Without Radiographic Progression in the Total Erosion Score at Week 104
Description: Total Erosion Score is determined by evaluation of fourteen sites in each wrist and hand and six joints in each foot using an eight-point scale from 0 (normal: no erosions) to 3.5 (Very severe; erosions of 100% of the articular surfaces. The score at baseline is compared to the score at week 104.
  No progression is defined as a change from score at screening to week 104 ≤0.
Time Frame: Week 104
Population: Participants from the Modified Intent to Treat (MITT) population includes all randomized participants who received at least one infusion and had both screening and post-baseline radiographic assessments. Patients with missing data are classified as progressing.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Number analyzed (Participants) | 233 | 239 | 244
Percentage of Participants | 38.2 | 52.7 | 58.6

30. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Week 104
Description: The Stanford Health Assessment Questionnaire disability index (HAQ-DI) is a patient completed questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. Each domain has at least two component questions. There are four possible responses for each component ranging from 0(without any difficulty) to 4 (unable to do). HAQ-DI=sum of worst scores in each domain divided by the number of domains answered. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 104
Population: Participants from the Intent-to treat Population includes all randomized participants who received at least one dose of study drug with data at baseline and Week 104 available for analysis. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Number analyzed (Participants) | 248 | 247 | 248
Score on a scale | -0.806 (0.7968) | -1038 (0.8142) | -1.055 (0.7901)
Statistical Analysis 1: Comparison: Placebo + Methotrexate vs Rituximab (0.5 g x 2) + Methotrexate; Rituximab (0.5 g x 2) + Methotrexate versus Placebo + Methotrexate, stratified for region and baseline RF status; Test type: Superiority or Other; p < 0.0001, ANOVA — Secondary endpoint in hierarchical testing structure
Statistical Analysis 2: Comparison: Placebo + Methotrexate vs Rituximab (1.0 g x 2) + Methotrexate; Rituximab (1.0 g x 2) + Methotrexate versus Placebo + Methotrexate, stratified for region and baseline RF status; Test type: Superiority or Other; p < 0.0001, ANOVA — Secondary endpoint in hierarchical testing structure

ADVERSE EVENTS:
Time Frame: From Baseline to End of ESFU
Description: Safety Population includes all participants who received at least one dose of study drug, grouped as treated. After Week 104 participants in the placebo group were eligible to receive either Rituximab 2 X 0.5 g + MTX or Rituximab 2 X 1.0g + MTX. Adverse events reported for placebo patients after switching to Rituximab are not included below.
Arm/Group | Placebo + Methotrexate | Rituximab (0.5 g x 2) + Methotrexate | Rituximab (1.0 g x 2) + Methotrexate
Serious Adverse Events (participants affected / at risk) | 48/249 | 54/348 | 58/263
Other Adverse Events (participants affected / at risk) | 193/249 | 232/348 | 208/263
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Methotrexate (N=249) | Rituximab (0.5 g x 2) + Methotrexate (N=348) | Rituximab (1.0 g x 2) + Methotrexate (N=263)
Pneumonia (Infections and infestations) | 6 | 7 | 4
Urinary Tract Infection (Infections and infestations) | 4 | 2 | 0
Appendicitis (Infections and infestations) | 0 | 2 | 0
Acute Tonsillitis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 1
Febrile Infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 1
Infection (Infections and infestations) | 0 | 0 | 3
Lung Infection (Infections and infestations) | 0 | 1 | 0
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 0 | 1 | 0
Pneumonia Pneumococcal (Infections and infestations) | 0 | 1 | 0
Septic Shock (Infections and infestations) | 0 | 1 | 0
Subcutaneous Abscess (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1 | 0
Appendicitis Perforated (Infections and infestations) | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Diverticular Perforation (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal Hypomotility (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal Hernia, Obstructive (Gastrointestinal disorders) | 0 | 1 | 1
Carotid Arteriosclerosis (Nervous system disorders) | 0 | 0 | 1
Embolic Stroke (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1 | 0
Carcinoma In Situ of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Primary Mediastinal Large B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 0 | 1
Surgical Failure (General disorders) | 0 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 2 | 1
Angina Pectoris (Cardiac disorders) | 1 | 0 | 0
Angina Unstable (Cardiac disorders) | 1 | 0 | 1
Atrioventricular Block Complete (Cardiac disorders) | 0 | 1 | 0
Angiopathy (Vascular disorders) | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0
Hypertensive Crisis (Vascular disorders) | 0 | 0 | 1
Pelvic Venous Thrombosis (Vascular disorders) | 1 | 0 | 0
Venous Insufficiency (Vascular disorders) | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 2 | 1
Accident (Injury, poisoning and procedural complications) | 1 | 0 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 2 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1
Calculus Urinary (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Vertigo Positional (Ear and labyrinth disorders) | 1 | 0 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 2
Cystocele (Reproductive system and breast disorders) | 0 | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 1
Metastatic Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Status Asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chest Pain (General disorders) | 1 | 2 | 2
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Endophthalmitis (Infections and infestations) | 0 | 1 | 0
Gangrene (Infections and infestations) | 1 | 0 | 0
Pulmonary Tuberculosis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Abdominal Hernia (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal Ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 1
Rectal Polyp (Gastrointestinal disorders) | 1 | 0 | 0
Umbilical Hernia (Gastrointestinal disorders) | 0 | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate Cancer Stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Intentional Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 2 | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 1 | 1
Hypertensive Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Laryngeal Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 2
Ulcer Haemorrhage (General disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0
Peripheral Ischaemia (Vascular disorders) | 0 | 1 | 0
Peripheral Vascular Disorder (Vascular disorders) | 0 | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Liver Disorder (Hepatobiliary disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Drug Dependence (Psychiatric disorders) | 0 | 1 | 0
Cervical Dysplasia (Reproductive system and breast disorders) | 2 | 0 | 0
Meniere's Disease (Ear and labyrinth disorders) | 1 | 0 | 0
Goitre (Endocrine disorders) | 1 | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Abortion Induced (Surgical and medical procedures) | 0 | 0 | 1
Pyelonephritis Acute (Infections and infestations) | 1 | 2 | 0
Dengue Fever (Infections and infestations) | 0 | 1 | 1
Abscess Limb (Infections and infestations) | 0 | 1 | 0
Arthritis Bacterial (Infections and infestations) | 0 | 0 | 1
Atypical Pneumonia (Infections and infestations) | 0 | 0 | 1
Colonic Abscess (Infections and infestations) | 0 | 1 | 0
H1N1 Influenza (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1
Necrotising Fasciitis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 1
Endometrial Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Anaplastic Large-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Monoclonal Gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Paget's Disease of Nipple (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colitis Ulcerative (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal Perforation (Gastrointestinal disorders) | 1 | 0 | 0
Large Intestinal Stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Multiple Fractures (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0
Coronary Artery Occlusion (Cardiac disorders) | 0 | 0 | 1
Mitral Valve Sclerosis (Cardiac disorders) | 0 | 0 | 1
Pericardial Effusion (Cardiac disorders) | 0 | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cereberal Infarction (Nervous system disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Ovarian Cyst Ruptured (Reproductive system and breast disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1
Diabetic Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1
Gastrointestinal Dysplasia (Gastrointestinal disorders) | 0 | 1 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cerebral Infarction (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Methotrexate (N=249) | Rituximab (0.5 g x 2) + Methotrexate (N=348) | Rituximab (1.0 g x 2) + Methotrexate (N=263)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 53 | 69 | 67
Nausea (Gastrointestinal disorders) | 42 | 45 | 46
Upper Respiratory Tract Infection (Infections and infestations) | 44 | 59 | 58
Nasopharyngitis (Infections and infestations) | 43 | 53 | 52
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 42 | 30 | 29
Urinary Tract Infection (Infections and infestations) | 26 | 36 | 43
Headache (Nervous system disorders) | 18 | 17 | 31
Anaemia (Blood and lymphatic system disorders) | 25 | 14 | 19
Hypertension (Vascular disorders) | 18 | 22 | 24
Diarrhoea (Gastrointestinal disorders) | 15 | 24 | 18
Bronchitis (Infections and infestations) | 15 | 32 | 20
Dizziness (Nervous system disorders) | 13 | 12 | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 19 | 24
Sinusitis (Infections and infestations) | 11 | 23 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 19 | 9
Pharyngitis (Infections and infestations) | 16 | 14 | 14
Dyspepsia (Gastrointestinal disorders) | 13 | 15 | 14
Gastritis (Gastrointestinal disorders) | 13 | 11 | 10
Gastroenteritis (Infections and infestations) | 7 | 9 | 16
Influenza (Infections and infestations) | 11 | 9 | 16
Drug-Induced Liver Injury (Hepatobiliary disorders) | 35 | 37 | 38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.